CLINICAL TRIAL: NCT06390215
Title: The School Readiness Journey: Capturing the Unheard Voices of Latino Parents
Brief Title: Clinic-Based School Readiness Coaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jaime Peterson, Assistant Professor of Pediatrics, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00021040; PPQ#1023820 (Other Grant/Funding Number: OHSU Health IDS, LLC)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: School Readiness
Keywords: School Readiness; Kindergarten; Early Learning; Coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School Readiness Coaching Intervention (Experimental): Two 1-hr individualized parent-child School Readiness Coaching Sessions conducted with Community Health Worker to assess child and parent school readiness skills and behaviors and provide parents with modeling, tools, and resources to support parent early math and literacy skills for home practice and connect them to preschool and community resources.
  Interventions: Behavioral: School Readiness Coaching Intervention

INTERVENTIONS:
Behavioral: School Readiness Coaching Intervention — Two 1-hr School Readiness Coaching Session

SUMMARY:
The goal of this clinical trial is to examine how a clinic-based school readiness coaching session conducted by a community health worker for parents of 3-5-year-olds affects children's School Readiness (SR) skills and parents early SR knowledge and behaviors. The main questions it aims to answer are: What impact does the clinic-based coaching session have on preschool-aged children's school readiness skills and their parents' confidence in supporting and practicing early math and literacy behaviors at home? Participants will receive a 1-hr coaching session at their pediatric clinic and return after three months for a follow-up session. Researchers will compare pre-and-post child and parent SR outcomes between these two sessions.

DETAILED DESCRIPTION:
The goal of this clinical trial is to examine how a clinic-based school readiness coaching session conducted by a community health worker for parents of 3-5-year-olds affects children's school readiness (SR) skills and parents early SR knowledge and behaviors. The main questions it aims to answer are: What impact does the clinic-based coaching session have on preschool-aged children's school readiness skills as measured by the Brigance Early Childhood Screen III? and What impact does the clinic-based coaching session have on parents' confidence in supporting and practicing early math and literacy behaviors at home using the DREME Parent Beliefs Survey? The secondary question this study aims to evaluate is: Does the 1-hr school readiness coaching session affect rates of well-child checks at the pediatric clinic? Participants will receive a 1-hr coaching session at their pediatric clinic and return after three months for a follow-up session. Researchers will compare pre-and-post Brigance scores for the child and pre-and post parent SR confidence DREME scores.

ELIGIBILITY:
Inclusion Criteria:

* Receives primary care at one of 2 clinic sites
* Parent or caregiver of 3-6-year-old
* Child is eligible for Medicaid services
* Parent and child can communicate in English or Spanish

Exclusion Criteria:

* Child is too ill to participate
* Parents who are unable to complete study activities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in child's school readiness skills measured by the Brigance Early Childhood Screen III for 3-5-year-olds. | Baseline and month 3
  The Early Childhood Screens III, available in three age-specific volumes, evaluate the key predictors of school success across the domains of Physical Development, Language Development, Academic Skills/Cognitive Development, and Self-help and Social-Emotional Skills. Composite score range is 0-100 with higher score indicating a better outcome.
Change in parent confidence teaching math and literacy measured by the DREME Parent Beliefs Survey | Baseline and month 3
  The DREME Parent Beliefs Survey is composed of 6 items that assess parent confidence and beliefs regarding teaching and practicing math and literacy with their child.

SECONDARY OUTCOMES:
Change in rates of well-child checks at the pediatric clinic. | Year one and year two
  Clinic will generate well-child checks reports for children enrolled to compare to clinic average.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Peterson, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No